CLINICAL TRIAL: NCT05336318
Title: Evaluation of a Peer Supported Program for Adolescent and Young Adult Cancer Patients
Brief Title: Peer2Me: A Peer Supported Program for Adolescent and Young Adult Cancer Patients
Acronym: Peer2Me
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Prof. Anja Mehnert-Theuerkauf, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DKH-70114047
Record Dates: First submitted 2022-02-04; First posted 2022-04-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Psychosocial Problem
Keywords: adolescents and young adulthood; AYA; psychooncology; peer-support
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Comprehensive cohort studies (CCS) are characterized by incorporating patient preferences into the study by using a "parallel preference group." The procedure is to ask patients' preferences at the beginning of the study before randomization. Those who do not consent to randomization will be retained in the study, but group assignment will be made according to their preferences. Patients who agree to randomization are randomized to one of the two groups (intervention vs. control).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Peer support
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Peer support — patients were supported by a mentor
  Arms: Intervention group

SUMMARY:
The present bicentric study has the aim to investigate the effectiveness of the peer supported mentoring program 'Peer2Me' with regard to psychosocial parameters using a prospective Comprehensive Cohort Design. Over a period of three months, acutely ill patients in the intervention group are accompanied by a mentor with the same disease and of similar age. Patients in the control group receive a one-time consultation. Before and after the intervention, mentors and mentees are interviewed about their psychosocial distress and quality of life.

DETAILED DESCRIPTION:
After successful piloting of the mentoring program "Peer2Me", the mentoring program developed by us is now to be implemented and evaluated in a large-scale study in a second step, in order to be able to derive clinically relevant results.

A total of 180 acutely ill adolescent and young cancer patients (AYA) between the ages of 18 and 39 will be included in the study (intervention and control group). Again, young former cancer patients who have completed treatment will act as mentors and accompany acutely ill AYAs in the period after diagnosis for a period of three months. Prior to their assignment, the mentors take part in a training course, which includes the teaching of suitable conversation techniques, core topics in dealing with the cancer and advice on further care structures. Patients in the control group receive 30 minutes of standardized counseling regarding psychosocial care needs, including appropriate informational materials, during AYA consultation hours at both clinic sites. The study includes three measurement time points: t1: before the intervention; t2: after the end of the intervention; t3: 3 months after the end of the intervention. At all time points, participants will be surveyed using standardized questionnaires. With the help of these data and a comprehensive statistical analysis, the investigators want to make valid statements regarding the effects of peer mentoring on changes in psychological well-being as well as on social support and coping with illness.

ELIGIBILITY:
Inclusion Criteria:

* Cancer disease between the ages of 18 and 39 (all tumor entities)
* completion of acute treatment at least 2 years ago (mentors)
* curative prognosis
* Native language German or fluent German speaker
* first cancer diagnosis in the last 6 months (mentees, all tumor entities)
* curative prognosis

Exclusion Criteria:

* existing and already diagnosed psychiatric disease, ongoing psychotherapy and/or existing suicidal tendency
* palliative treatment approach

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessing post traumatic growth of mentors and change | Baseline and 3 months after intervention
  The Posttraumatic Growth Inventory (PTGI) measures the extent to which patients have experienced positive changes regarding cancer. The questionnaire contains 21 items in the five dimensions: new opportunities, relationship with others, personal strength, appreciation of life, and spiritual change. Using a three-point Likert scale, patients indicate the extent to which the item responses apply. Item scores are summed to form a total score, with higher scores indicating higher posttraumatic growth.
Assessing Empathy of mentors and change | Baseline and 3 months after intervention
  The Saarbrücken Personality Questionnaire on Empathy is the German adaptation of the Interpersonal Reactivity Index. The SPF is a questionnaire for self-assessment of one's own empathic abilities and consists of 16 items that measure both the cognitive and the emotional dimension of empathy on four subscales: imagination, empathic distress, empathic sympathy, and perspective taking.
  A five-point Likert scale (1- never to 5- always) is used to assess the extent to which the statements are true.
Life satisfaction of mentors and change | Baseline and 3 months after intervention
  The FLZ-M is a valid instrument that measures the subjective assessment of satisfaction in various areas of life. Life satisfaction is assessed using the two modules "general life satisfaction" and "satisfaction with health", each with eight items and one overall item. Subjective satisfaction and importance are assessed on a five-point Likert scale (0 = "dissatisfied" to 4 = "very satisfied").
Life satisfaction of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  The FLZ-M is a valid instrument that measures the subjective assessment of satisfaction in various areas of life. Life satisfaction is assessed using the two modules "general life satisfaction" and "satisfaction with health", each with eight items and one overall item. Subjective satisfaction and importance are assessed on a five-point Likert scale (0 = "dissatisfied" to 4 = "very satisfied").
Self-efficacy of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  The General Self-Efficacy Expectancy Scale is a self-assessment procedure with 10 items for assessing general optimistic self-convictions. It measures the expectation of subjective competence to cope with difficult situations such as cancer.
  A four-point Likert scale is used to ascertain the extent to which patients agree with the statements. The individual test score is calculated by summing up all ten items.
Coping of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  Self-efficacy in coping with cancer can be defined as the confidence of a cancer patient in his or her ability to develop adaptive coping behavior. The German version of the short form of the Cancer Behavior Inventory (CBI-B-D) uses 14 items to describe coping behavior in the context of cancer. Patients estimate on a nine-point Likert scale how confident they are in performing certain behaviors. By summing all 14 item scores, a sum score is obtained, with high scores indicating high confidence in the ability to perform the coping behavior.
Anxiety of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  The Generalized Anxiety Scale measures symptoms of generalized anxiety disorders and the symptom severity of generalized anxiety on a four-point Likert scale using seven items. The individual item scores are summed to a total score, which can assume values between 0 and 21 points.
Depressive symptoms of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  The Patient Health Questionnaire measures depressive symptoms on a four-point Likert scale using nine items. The PHQ-9 can be evaluated both categorically and by summing up the item characteristics. The scale sum value can reach values between 1 and 27.
Social support of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  The Berlin Social Support Scales measure six dimensions of social support in a multidimensional approach: perceived social support, received social support, provided social support, need and search for social support, and protective cushioning in the sense of protecting others from stress.
Health literacy of mentees and change | Baseline and 3 months after intervention and 6 months after intervention
  The HLS-EU-Q16 measures health literacy with 16 items and was developed from the long version of the HLS-EU-Q47. The items refer to various tasks and activities related to health care, disease prevention or health promotion. Respondents rate in each case how easy they think the corresponding task or activity is ("very easy," "fairly easy," "fairly difficult," "very difficult"). A sum score from 0 to 16 can be calculated, and the latter can be classified as insufficient (<9), problematic (9-12), and sufficient (13-16) health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Richter, PhD., Principal Investigator — Universitätsklinikum Leipzig; Corinna Bergelt, Prof., Principal Investigator — University Medicine Greifswald, Institute for Medical Psychology
Locations (2):
- Germany (2):
  - University Medical Center Leipzig, Leipzig, Saxony
  - University Medical Center Hamburg-Eppendorf, Department of Medical Psychology, Hamburg

REFERENCES:
- [Derived] Brock H, Dwinger S, Friedrich M, Sender A, Geue K, Mehnert-Theuerkauf A, Bergelt C, Richter D. Peer2Me - impact of peer support on self-efficacy in young adult cancer survivors (YA-CS): findings from a comprehensive cohort design. BMC Cancer. 2025 May 26;25(1):943. doi: 10.1186/s12885-025-14323-5. PMID 40420294
- [Derived] Brock H, Dwinger S, Bergelt C, Sender A, Geue K, Mehnert-Theuerkauf A, Richter D. Peer2Me - evaluation of a peer supported program for adolescent and young adult (AYA) cancer patients: study protocol of a randomised trial using a comprehensive cohort design. BMC Cancer. 2024 Jul 2;24(1):788. doi: 10.1186/s12885-024-12547-5. PMID 38956510